CLINICAL TRIAL: NCT03431025
Title: Wrist-worn Sensors for Tele-Rehabilitation of the Hemiparetic Upper Extremity; A Feasibility Study
Brief Title: Wrist-worn Sensors for Tele-Rehabilitation of the Hemiparetic Upper Extremity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BioSensics (Industry)
Collaborators: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P001688/SRH
Record Dates: First submitted 2018-01-23; First posted 2018-02-13 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Stroke; Hemiparesis
MeSH Terms: conditions — Stroke; Paresis | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the Control Arm will wear sensors to monitor their upper limb movement but will not receive feedback from these sensors to encourage usage of the impaired limb during activities of daily living.
- Intervention (Experimental): Participants in the Experimental Arm will wear sensors to monitor their upper limb movement and will receive feedback from these sensors to encourage usage of the impaired limb during activities of daily living.
  Interventions: Device: Wearable sensors and biofeedback

INTERVENTIONS:
Device: Wearable sensors and biofeedback — Participants in the Experimental Arm will wear sensors to monitor their upper limb movement and will receive feedback from these sensors to encourage usage of the impaired limb during activities of daily living.
  Arms: Intervention

SUMMARY:
Stroke and other causes of central nervous system damage can result in debilitating loss of motor control that is often more pronounced in one limb than the other. Using or attempting to use the affected limb during activities of daily living, despite considerable difficulty, stimulates neuroplasticity and motor function recovery. The investigators are conducting a clinical study to test the efficacy of wrist-worn sensors that encourage affected limb use during activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke at least 3 months prior to study enrollment
* Mild-to-moderate to severe upper-limb motor impairments (as measured by a score between 21 and 50 on the arm section of the Fugl-Meyer scale).

Exclusion Criteria:

* Cognitive impairments that would significantly interfere with their ability to follow instructions (as measured by a score lower than 23 on the Mini Mental State Examination scale)
* Severe attention deficits or hemispatial neglect (as measured by the Mesulam Cancellation test and the Line Bisection test);
* Severe range-of-motion limitations (as measured via physical examination) or severe spasticity (as measured using the Modified Ashworth scale) that would prevent safe performance of home-based exercises;
* Proprioceptive deficits that impair their ability to process feedback (as measured using the Fugl-Meyer Assessment-upper extremity; sensory section).
* Implantable medical devices that are not compliant with the ISO 14117:2012 and/or ANSI/AAMI PC69 standards for Bluetooth compatibility. We will ask subjects to provide us with their medical device record card and verify that the device complies with the above-mentioned standards. If not, they will be excluded from the study.
* Participation in upper-extremity rehabilitation program (i.e. outpatient occupational therapy, research study, ...).
* Recent (< 3 months) Botox injection in the upper-extremity or plan to undergo injections during the study timeline.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer during intervention | 12 weeks
  Change in Fugl-Meyer Upper Extremity Assessment Scale score from baseline (measure of upper extremity impairment, score range from 0 to 66 points, higher values are considered a better outcome).
Change in Motor Activity Log Quality Score during intervention | 12 weeks
  Change in Motor Activity Log Quality Score from baseline (measure of hemiparetic upper extremity use in daily life, score range from 0 to 5 points, higher values are considered a better outcome)
Change in Motor Activity Log Quantity Score during intervention | 12 weeks
  Change in Motor Activity Log Quantity Score from baseline (measure of hemiparetic upper extremity use in daily life, score range from 0 to 5 points, higher values are considered a better outcome)
Change in Fugl-Meyer during washout | 12 weeks (end of intervention), 20 weeks (follow-up)
  Change in Fugl-Meyer Upper Extremity Assessment Scale score from end of intervention to follow-up (measure of upper extremity impairment, score range from 0 to 66 points, higher values are considered a better outcome).
Change in Motor Activity Log Quality Score during washout | 12 weeks (end of intervention), 20 weeks (follow-up)
  Change in Motor Activity Log Quality Score from end of intervention to follow-up (measure of hemiparetic upper extremity use in daily life, score range from 0 to 5 points, higher values are considered a better outcome)
Change in Motor Activity Log Quantity Score during washout | 12 weeks (end of intervention), 20 weeks (follow-up)
  Change in Motor Activity Log Quantity Score from end of intervention to follow-up (measure of hemiparetic upper extremity use in daily life, score range from 0 to 5 points, higher values are considered a better outcome)

SECONDARY OUTCOMES:
Change in Wolf Motor Function Test time-subscale during intervention | 12 weeks
  Change in Wolf Motor Function Test time-subscale score from baseline (measure of upper extremity function, score range from 0 to 120 seconds, lower values are considered a better outcome)
Change in Wolf Motor Function Test quality-subscale during intervention | 12 weeks
  Change in Wolf Motor Function Test quality-subscale score from baseline (measure of upper extremity function, score range from 0 to 5 points, higher values are considered a better outcome)
Change in Wolf Motor Function Test time-subscale during washout | 12 weeks (end of intervention), 20 weeks (follow-up)
  Change in Wolf Motor Function Test time-subscale score from end of intervention to follow-up (measure of upper extremity function, score range from 0 to 120 seconds, lower values are considered a better outcome)
Change in Wolf Motor Function Test quality-subscale during washout | 12 weeks (end of intervention), 20 weeks (follow-up)
  Change in Wolf Motor Function Test quality-subscale score from end of intervention to follow-up (measure of upper extremity function, score range from 0 to 5 points, higher values are considered a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph T Gwin, PhD, Principal Investigator — BioSensics; Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No